CLINICAL TRIAL: NCT06995183
Title: Improved Assessment of Cardiovascular Risk Through Imaging in Relatives Identified By Lipoprotein(a) Cascade Screening
Brief Title: Heart CT Imaging to Detect Early Coronary Artery Disease in First-Degree Relatives With High or Low Lipoprotein(a) Identified Through Family Screening
Acronym: IMAGE-LPA
Status: Recruiting | Type: Observational
Sponsor: E.S.stroes (Other)
Responsible Party: Sponsor-Investigator, E.S.stroes, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 2024.1104
Record Dates: First submitted 2025-05-16; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lipoprotein(a)
Keywords: Lipoprotein(a); coronary atherosclerosis; subclinical atherosclerosis; coronary artery calcium scoring; coronary computed tomography angiography; cardiovascular risk assessment; primary prevention; coronary artery disease; cascade screening; imaging biomarkers; atherosclerotic cardiovascular disease; lipid disorders
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Lp(a): Individuals aged 50 years or older who were identified with elevated Lipoprotein(a) levels (≥150 nmol/L) through familial cascade screening at the Amsterdam UMC Vascular Medicine outpatient clinic. These participants have no history of clinical atherosclerotic cardiovascular disease and are undergoing imaging to assess subclinical coronary atherosclerosis.
- Low Lp(a): Age- and sex-matched individuals aged 50 years or older with normal Lipoprotein(a) levels (<50 nmol/L), identified through the same familial cascade screening program. These participants also have no history of clinical atherosclerotic cardiovascular disease and serve as controls to compare the prevalence of subclinical coronary plaque.

SUMMARY:
Lipoprotein(a), or Lp(a), is a type of cholesterol that can increase the risk of heart and blood vessel disease. Many people are unaware they have high Lp(a), since it is not routinely measured and usually causes no symptoms on its own. However, elevated Lp(a) levels tend to run in families, meaning that close relatives of individuals with high Lp(a) are more likely to have it as well.

At Amsterdam UMC, family members of patients with high Lp(a) are invited for cascade screening, which includes testing for Lp(a) and other cardiovascular risk factors. From this screened group, a selection of individuals with either high or low Lp(a) levels are invited to participate in the IMAGE-LPA study.

In IMAGE-LPA, participants undergo a comprehensive cardiovascular evaluation, including blood tests and heart imaging using CT scans. Two types of scans are performed: (1) a calcium score scan to detect early calcium buildup in the heart's arteries (an early marker of atherosclerosis), and (2) coronary CT angiography to assess for plaque and narrowing in the coronary arteries.

The goal of the study is to compare individuals with high versus low Lp(a) identified through cascade screening, to determine whether high Lp(a) levels are associated with early signs of heart disease in this patient group.

The study does not involve any medications or invasive procedures. The findings may help clarify whether heart imaging can improve early detection in individuals with high Lp(a), and guide future strategies for preventing cardiovascular disease in families affected by this inherited risk factor.

ELIGIBILITY:
In order to be eligible to participate in this study in the elevated Lp(a) subgroup, a subject must meet all of the following inclusion criteria:

* Man or woman ≥50 years of age;
* Lp(a) level ≥ 150 nmol/L;
* Identified as having elevated Lp(a) through Lp(a) family cascade screening at the Amsterdam UMC Vascular Medicine outpatient clinic;
* Able and willing to provide informed consent;
* Able to comply with study requirements.

In order to be eligible to participate in this study in the Low Lp(a) subgroup, a subject must meet all of the following inclusion criteria:

* Man or woman ≥50 years of age;
* Lp(a) level < 50 nmol/L;
* Identified as having elevated Lp(a) through Lp(a) family cascade screening at the Amsterdam UMC Vascular Medicine outpatient clinic;
* Able and willing to provide informed consent;
* Able to comply with study requirements.

A potential subject who meets any of the following criteria will be excluded from participation in this study (both subgroups):

* Renal insufficiency, defined as eGFR < 30 ml/min
* History of ASCVD (acute coronary syndrome, history of myocardial infarction, stable or unstable angina pectoris or coronary or other arterial revascularization, stroke, transient ischemic attack or peripheral artery disease including aortic aneurysm, all of atherosclerotic origin)
* History of atrial fibrillation
* Prior and current use of statins
* Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
* Unable or unwilling to provide informed consent
* Unable to comply with study requirements.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from first-degree relatives of patients with elevated Lipoprotein(a) who previously participated in the Lp(a) familial cascade screening program at the Amsterdam UMC Vascular Medicine outpatient clinic. All participants have been screened for Lp(a) levels as part of routine clinical care and have indicated willingness to be contacted for future research. Eligible individuals are middle-aged or older and have no history of clinically manifest atherosclerotic cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Coronary Atherosclerotic Plaque Detected on CCTA | Day 1
  Assessment of the presence or absence of any coronary artery plaque as detected by coronary computed tomography angiography (CCTA). Plaque is defined as within and/or adjacent to the vessel lumen distinguishable from the lumen and surrounding tissue.

SECONDARY OUTCOMES:
Number of Participants with Obstructive Coronary Stenosis (≥50% Luminal Narrowing) on CCTA | Day 1
  Measured by CCTA. Obstructive stenosis is defined as luminal narrowing of ≥50% in any major coronary artery, based on visual assessment and automated quantification.
Total Coronary Plaque Volume | Day 1
  Total plaque volume (in mm³) across all coronary segments, quantified using FDA-approved software (Cleerly Inc.) from CCTA scans. Includes both calcified and non-calcified plaque.
Calcified and Non-Calcified Plaque Volumes | Day 1
  Volumes (in mm³) of calcified and non-calcified coronary plaque separately measured using semi-automated quantification of CCTA images. Non-calcified plaque includes fibrous and lipid-rich components.
Low-Attenuation Plaque Volume | Day 1
  Volume (in mm³) of coronary plaque with CT attenuation <30 HU, measured on CCTA. Low-attenuation plaque is associated with high-risk morphology and vulnerability.
Pericoronary Adipose Tissue (PCAT) Attenuation | Day 1
  Mean CT attenuation (in Hounsfield Units) of adipose tissue surrounding coronary arteries, as a surrogate of coronary inflammation. Measured on CCTA at the proximal right coronary artery.
Number of High-Risk Plaque Features | Day 1
  CCTA-based count of high-risk plaque features per patient, including positive remodeling, napkin-ring sign, low-attenuation plaque, and spotty calcification. A higher count suggests greater risk of future events.
Coronary Artery Calcium (CAC) Score | Day 1
  Agatston CAC score obtained from non-contrast CT scan preceding CCTA. Score quantifies coronary calcification.
  Scale: 0-400+; higher score = more calcification, worse outcome
CAD-RADS Classification | Day 1
  Coronary Artery Disease Reporting and Data System (CAD-RADS) score, a standardized grading system for coronary stenosis severity based on CCTA. Scores range from 0 (no plaque) to 5 (severe stenosis ≥70%).

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because participants did not provide explicit consent for their data to be shared beyond the scope of the approved study. Data sharing was not included as part of the informed consent process.

REFERENCES:
- [Background] Annink ME, Janssen ES, Reeskamp LF. Effectiveness of cascade screening for elevated lipoprotein(a), an underdiagnosed family disorder. Curr Opin Lipidol. 2024 Dec 1;35(6):290-296. doi: 10.1097/MOL.0000000000000951. Epub 2024 Sep 18. PMID 39259684